CLINICAL TRIAL: NCT03227770
Title: A Randomized, Open-label, Multi-centre Trial Comparing Hemodialysis Plus Hemoperfusion Versus Hemodialysis Alone in Adult Patients With End-stage Renal Disease (HD/HPvsHD)
Brief Title: The Benefit of Hemodialysis Plus Hemoperfusion on Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); RenJi Hospital (Other); Ruijin Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai 6th People's Hospital (Other); Changhai Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai University of Traditional Chinese Medicine (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Principal Investigator, Gengru Jiang, Director of Renal Division, Department of Internal Medicine, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-017
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: End-stage Renal Disease
Keywords: Hemoperfusion; Hemodialysis; Mortality
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular hemodialysis (Active Comparator): Blood purification (including low-flux hemodialysis, high-flux hemodialysis, or hemodiafiltration) treatment ≥10 hours per week
  Interventions: Device: hemodialysis
- hemoperfusion combined with hemodialysis (Experimental): Combination of hemodialysis and hemoperfusion treatment at least once every two week
  Interventions: Device: hemoperfusion combined with hemodialysis; Device: hemodialysis

INTERVENTIONS:
Device: hemoperfusion combined with hemodialysis — Hemoperfusion combined with hemodialysis treatment will perform at least once every two week. The hemoperfusion apparatus will use type HA130 resin hemoperfusion apparatus (Zhuhai Jafron Biomedical Co., Ltd, China)
  Arms: hemoperfusion combined with hemodialysis
Device: hemodialysis — Blood purification (including low-flux hemodialysis, high-flux hemodialysis, or hemodiafiltration) treatment ≥10 hours per week

SUMMARY:
This multi-center, open-label, randomized controlled trial aims to investigate the efficacy of hemoperfusion (HP) combined with hemodialysis (HD) by evaluating all-cause mortality and cardiovascular mortality in maintenance hemodialysis patients.

DETAILED DESCRIPTION:
In this HD/HPvsHD trial, we plan to enroll 1364 maintenance hemodialysis patients. Eleven medical centers in Shanghai Metropolitan area have explicitly expressed interest to participate. Participants will be randomized to receive hemodialysis plus hemoperfusion or hemodialysis alone at a 1:1 ratio after 1-month run-in period. In both arms, patients will receive lBlood purification (including low-flux hemodialysis, high-flux hemodialysis, or hemodiafiltration) treatment at least 10 hours per week. In the experiment group, in addition to the treatments in the control arm, hemoperfusion will be conducted at least once every two weeks using a HA130 resin hemoperfusion apparatus containing 130ml resin. Follow-up is scheduled at 3, 6, 12, 18, 24 and up to 48 months after randomization, and will consist the following: routine physical examinations, standard lab panels (blood routine, liver/kidney functions, tests of the coagulation system, etc.), chest X-ray, electrocardiogram, echocardiography, heart function rating (based on New York Heart Association grading). Dialysis adequacy defined by standard Kt/V will be calculated. Adverse events will be assessed according to the international conference on harmonization guidelines. The primary outcomes will include 24-month all-cause mortality. Secondary outcomes will include cardiovascular-related mortality, the occurrence of major cardiovascular events and the quality of life (Kidney Disease Quality of Life Short Form).

ELIGIBILITY:
Patients must meet all of the following criteria are eligible:

1. Age ≥ 18 years old
2. Regular blood purification treatment at least 3 months before enrolled in this study

3) Standard Kt/V ≥ 1.2

Subjects with one of more of the following conditions will be excluded:

1. White blood cell count < 4×10^9/L and / or platelet count < 100×10^9/L
2. Cerebral hemorrhage in the past 12 weeks
3. MACEs in the past 8 weeks
4. Severe heart failure (New York Heart Association [NYHA] class IV)
5. Active gastrointestinal bleeding, or coagulation dysfunction
6. Malignant tumor
7. Active infection
8. Pregnancy or lactation 9) Mental disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1362 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | From date of enrollment until the end of study, assessed up to 24 months
  Compared the difference between standardized therapy and hemoperfusion combined with hemodialysis treatment

SECONDARY OUTCOMES:
Cardiovascular-related mortality and major cardiovascular events (MACEs) | From date of enrollment until the end of study, assessed up to 24 months
  Major cardiovascular events events including angina pectoris, acute myocardial infarction, severe arrhythmia, congestive heart failure, myocarditis, pericarditis, cardiac surgery or peripheral vascular surgery, stroke and peripheral vascular disease
Evaluation of quality of life | From date of enrollment until the end of study, assessed up to 24 months
  Assessment of quality of life using the KDQOL-SF (Kidney Disease Quality of Life Short Form) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gengru Jiang, doctoral, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (11):
- China (11):
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Yangpu District Central Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
The mortality data will be shared

REFERENCES:
- [Derived] Lu W, Jiang GR; HD/HP versus HD trial Group. Randomised, open-label, multicentre trial comparing haemodialysis plus haemoperfusion versus haemodialysis alone in adult patients with end-stage renal disease (HD/HP vs HD): study protocol. BMJ Open. 2018 Jul 28;8(7):e022169. doi: 10.1136/bmjopen-2018-022169. PMID 30056391

DOCUMENTS (1):
  • Study Protocol (2018-04-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT03227770/Prot_002.pdf